CLINICAL TRIAL: NCT05911048
Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant COVID-19 Bivalent (XBB+Prototype) Protein Vaccine (Sf9 Cell) (WSK-V101C) in Booster Vaccination in Healthy Population 18 Years Old of Age and Above
Brief Title: A Clinical Trial of Recombinant COVID-19 Bivalent (XBB+Prototype) Protein Vaccine (Sf9 Cell) in Booster Vaccination
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WSKCT016
Record Dates: First submitted 2023-06-16; First posted 2023-06-20 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Recombinant COVID-19 Bivalent (XBB+Prototype) Protein Vaccine (Sf9 Cell) (WSK-V101C)
  Interventions: Biological: Recombinant COVID-19 Bivalent (XBB+Prototype) Protein Vaccine (Sf9 Cell) (WSK-V101C)
- Control group (Active Comparator): Recombinant COVID-19 Vaccine (Sf9 Cell)(WSK-V101)
  Interventions: Biological: Recombinant COVID-19 vaccine(Sf9 Cell) (WSK-V101)

INTERVENTIONS:
Biological: Recombinant COVID-19 Bivalent (XBB+Prototype) Protein Vaccine (Sf9 Cell) (WSK-V101C) — boost with Recombinant COVID-19 Bivalent (XBB+Prototype) Protein Vaccine (Sf9 Cell) (WSK-V101C)
  Arms: Experimental group
Biological: Recombinant COVID-19 vaccine(Sf9 Cell) (WSK-V101) — boost with Recombinant COVID-19 vaccine (Sf9 Cell) (WSK-V101)
  Arms: Control group

SUMMARY:
A Clinical Trial of Recombinant COVID-19 Bivalent (XBB+Prototype) Protein Vaccine (Sf9 Cell) in Booster Vaccination to evaluate safety and immunogenicity in healthy population aged 18 years old and above.

DETAILED DESCRIPTION:
To evaluate safety of Recombinant COVID-19 Bivalent (XBB+Prototype) Protein Vaccine (Sf9 Cell) (WSK-V101C) and immunogenicity superiority of WSK-V101C to Recombinant COVID-19 vaccine (WSK-V101) after booster.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years and above, including those with underlying diseases and immunocompromised subjects.
2. Basic or booster immunization with COVID-19 vaccine ≥6 months.
3. ≥3 months of SARS-CoV-2 infection history, or never infected.
4. Have the ability to understand research procedures, with informed consent, voluntarily sign informed consent, and be able to comply with the requirements of clinical research protocols.

Exclusion Criteria:

1. Axillary temperature ≥37.3℃.
2. SARS-CoV-2 antigen or nucleic acid screening positive within the last 48 hours.
3. Anti-SARS-CoV-2 IgM antibody was positive during the screening period.
4. It is in the advanced stage of malignant tumor and the disease control is unstable.
5. Female pregnancy (pregnancy test results are positive), lactation period.
6. Have serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, heart failure, severe hypertension, and can not be controlled by drugs.
7. Have other serious chronic conditions such as uncontrolled asthma, diabetes, chronic obstructive pulmonary disease, pulmonary embolism, chronic kidney disease requiring dialysis, cirrhosis of the liver, convulsions, epilepsy and other neurological/psychiatric conditions.
8. Have been diagnosed with congenital or acquired immunodeficiency, HIV infection.
9. People who are allergic to any component of the investigational vaccine have a history of more severe allergies or allergic reactions to the vaccine in the past.
10. Congenital or acquired angioedema/neuroedema.
11. Asplenia or functional asplenia.
12. Thrombocytopenia or other clotting disorders (which may cause intramuscular injection contraindications).
13. Received another investigational drug within 1 month prior to receiving the investigational vaccine.
14. Received subunit or inactivated vaccine within 14 days prior to receiving the investigational vaccine, or received live attenuated vaccine within 1 month.
15. Fertile female subjects did not use effective contraception within 1 month prior to enrollment.
16. Fertile female and male subjects have pregnancy plans and sperm/egg donation plans from the screening period to 3 months after immunization.
17. Abnormal laboratory test results during the screening period, which were judged by the researcher to be unsuitable for the study vaccine.
18. Medical, psychological, social, or other conditions that, in the investigator's judgment, are inconsistent with the protocol or affect the subject's signing of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3100 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
AE and AR | 0-7 days after vaccination
  Incidence of adverse events (AE) and adverse reactions (AR) 0-7 days after vaccination.
Primary Immunogenicity indicator | day 14 post-vaccination
  The geometric mean titer (GMT) and seroconversion of neutralizing antibodies (true virus or pseudovirus method) against the current variants of SARS-CoV-2 (such as XBB and its subtypes) at day 14 post-vaccination.

SECONDARY OUTCOMES:
AE and AR | 0-30 days post-vaccination.
  Incidence of adverse events (AE) and adverse reactions (AR) 0-30 days post-vaccination.
SAE and AE | within12 months post-vaccination.
  Incidence of serious adverse events (SAE) and adverse events of specific interest (AESI) within 12 months post-vaccination.
Secondary Immunogenicity indicator 1 | day 14 post-vaccination.
  Geometric mean titer (GMT) and seroconversion rate of neutralizing antibody (true virus or pseudovirus method) against SARS-CoV-2 prototype strain and Omicron BA.2 variant strain on day 14 post-vaccination.
Secondary Immunogenicity indicator 2 | day 14 post-vaccination
  Geometric mean fold increase (GMI) of neutralizing antibodies against SARS-CoV-2 prototype strains, current variants (such as XBB and its subtypes), and Omicron BA.2 variants (true virus or pseudovirus method) on day 14 post-vaccination.
Secondary Immunogenicity indicator 3 | day 30 post-vaccination.
  Geometric mean titer (GMT), seroconversion rate and geometric mean fold increase (GMI) against SARS-CoV-2 prototype strains, current variants (such as XBB and its subtypes) and Omicron BA.2 variants neutralizing antibodies (true virus or pseudovirus method) at day 30 post-vaccination.
Secondary Immunogenicity indicator 4 | 14 and 30 days post-vaccination.
  Geometric mean titer (GMT), seroconversion rate and geometric mean fold increase (GMI) of anti-SARS-CoV-2 specific binding antibodies at 14 and 30 days after vaccination.